CLINICAL TRIAL: NCT06076577
Title: Does a Pre-operative Exercise Program Improve Post-operative Outcomes in Patients Undergoing Spinal Fusion Surgery for Adolescent Idiopathic Scoliosis?
Brief Title: Does a Pre-operative Exercise Program Improve Post-operative Outcomes for Fusion Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Firoz Miyanji, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H22-02186
Record Dates: First submitted 2023-04-24; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention)
- Prehabilitation Exercise Group (Experimental): The exercise arm participants will be asked to complete weekly questionnaires which will take around 10 minutes each week and the exercise program which takes 30 minutes each day.
  Interventions: Behavioral: Prehabilitation Exercise Group

INTERVENTIONS:
Behavioral: Prehabilitation Exercise Group — A set of core stabilization exercises and scoliosis specific exercises will be given to patients.
  Arms: Prehabilitation Exercise Group

SUMMARY:
A study found that in 1744 patients undergoing fusion surgery for adolescent Idiopathic scoliosis, 12% had back pain remaining after recovering from surgery. Rehabilitation prior to spine surgery or prehabilitation (prehab), has been shown to reduce costs and improve functional outcomes in patients who have had total hip or total knee arthroplasties. There is a lack of literature looking at prehab in the context of spine surgeries. The purpose of this study is to see if prehab can improve patient outcomes such as decreased pain, decreased length of stay in the hospital, and improved functional outcomes in patients undergoing fusion surgery for adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is the most common spinal deformity in adolescents and literature suggests that the link between back pain and AIS is underreported. Core stabilization exercises and scoliosis specific exercises have been shown to increase SRS scores related to pain (higher SRS scores indicate lower levels of pain). Additionally, higher SRS scores at pre-op were associated with a lower risk of residual postoperative pain following a fusion surgery. This suggests that preoperative exercise programs should lead to an increase in SRS pain scores post-operatively however, this direct relationship has not been researched. Rehabilitation exercises prior to surgery has been shown to improve functional outcomes in knee and hip arthroplasties however, the rehabilitation preoperatively has not been studies in the context of spine surgeries. The purpose of this study is to evaluate whether the prehabilitation exercise program can improve post-op outcomes including length of stay, decreased pain, decreased length of stay, and improved functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Included patients will have a diagnosis of AIS (ages 11-18). They will have a curve angle requiring surgery and be on the waitlist for surgery.

Exclusion Criteria:

* Patients will be excluded if they are currently enrolled in a physiotherapy designed exercise program prior to being enrolled in the study.
* They will be excluded if they have additional medical issues, limiting their ability to participate fully in the exercise program.
* Individuals with any cognitive disability that affects their ability to complete the questionnaires or follow instructions for the exercise program will also be excluded.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 2 years
  The primary analysis for the primary outcome length of stay is to determine if the prehab program reduces the average length of stay. It will follow the intention to treat approach, which will include all randomized participants retained in the group to which they are allocated. A complete analysis will be conducted to compare the outcomes between the two arms, utilizing the Student's t test or Wilcoxon-Mann-Whitney test, as appropriate for the distribution of the data. If more than 10% of randomized participants have missing length of stay outcomes, the missing data will be imputed using the Last Observation Carried Forward approach, as a sensitivity analysis.

SECONDARY OUTCOMES:
Pain Outcome | 2 years
  The pain outcomes will be measured using the Visual Analogue Scale (VAS); a scale ranging from 0 - 10, where 0 indicates no pain, and 10 indicates extreme pain.
Functional Outcome | 2 years
  The functional outcomes will be measured using the Scoliosis Research Society 22-item questionnaire (SRS-22). In this questionnaire, responses correspond to numbers 1 - 5, where 1 is the worst possible outcome and 5 is the best possible outcome. There will be a total SRS-22 score (average of all the scores) and five sub scores. The sub scores will be divided into five groups: function, pain, self-image, mental health, and satisfaction with management. Answers to questions relating to these categories will be averaged for each sub score.

IPD SHARING:
Plan to Share IPD: No